CLINICAL TRIAL: NCT02430792
Title: Effectiveness of Community-based Football Compared With Usual Care on Quality of Life in Men With Prostate Cancer: the FC Prostate Community Randomized Controlled Trial
Brief Title: Effectiveness of Community-based Football in Prostate Cancer
Acronym: FC-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: TrygFonden, Denmark (Industry); University of Copenhagen (Other); Parker Research Institute (Other); The Danish Football Association (Unknown); Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Eik Bjerre, Msc. PhD. Student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IDnr. 106471
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Prostate Cancer
Keywords: Prostatic Neoplasms; Exercise; Football; Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Football (Active Comparator): Recreational football 1-hour twice weekly in a local football club on a disease specific team
  Interventions: Behavioral: Football
- Control (No Intervention): A 15-30-minute guidance session upon group allocation to encourage engagement in the standard rehabilitation offered by the municipality

INTERVENTIONS:
Behavioral: Football — The football training will consist of sessions of 20 minutes of warm-up exercises. Followed by 20 minutes dribbling, passing, shooting exercises. Ends with 20 minutes of 5-7 a-side games.
  Arms: Football

SUMMARY:
Prostate cancer is the most common malignancy in men. Three million are currently living in the United States with the disease and this number is expected to rise to four million in 2024. Most live many years with the disease and experience significant morbidity both due to disease progression and treatment toxicity. Exercise has shown to improve QoL and reduce treatment toxicity. Moreover epidemiological evidence has suggested that physical activity improves survival.

Football has been shown to induce positive effects on body composition and bone markers in a subgroup of prostate cancer patients, those receiving androgen deprivation therapy.

The objective is to examine the effectiveness of football in prostate cancer survivors.

DETAILED DESCRIPTION:
PLAN FOR THE STATISTICAL ANALYSES

This plan has been prepared and is laid forward before any follow-ups are conducted. The plan delineates the analyses of the FC PC trial; any deviations will be laid forward and discussed in the final publication.

The primary statistical analysis targets the effect on prostate cancer (PCa) specific Quality of Life (QoL) of a treatment policy offering community based football to men with prostate cancer. In particular, patients will be analysed in the treatment group to which they were randomly allocated respecting the intention-to-treat principle (ITT). The appropriate method for addressing this effect depends on the assumptions made about missing data (drop-outs). Our main analysis is valid under the missing at random assumption but we will also present sensitivity analyses robust to non-ignorable patterns among patients with incomplete data.

Per protocol analyses will be performed to estimate the de jure effect of the treatment for compliant patients. The "per protocol" population will be defined as those trial participants from the intervention group that have attended the football intervention at least 12 times in the first 12 weeks and 24 times in 6 months intervention period.

Significance tests will be two-sided with a maximal type I error risk of 5 %. To address the problem of multiple comparisons for secondary analyses when several outcomes are tested or multiple constracts are extracted from the same statistical model p-values will be adjusted using the step-down Bonferrroni method of Holm (Holm 1979) or appropriate modern alternatives.

Trial profile A CONSORT diagram will show trial participant flow. Number of screened patients fulfilling inclusion criteria and trial subjects included in analyses together with reasons for exclusion of trial subjects will be reported.

Primary outcome The continuous outcome score of FACT-P will be calculated using the official scoring guideline. As described in the scoring guideline missing items will be prorated by multiplying the sum of the subscale with the number of the items in the subscale, then divided by the number of items answered. This will only be done if more than 50% of the items are answered in the subscales and 80% are answered in the total questionnaire. The change score of the total FACT-P at 12 weeks will be calculated by subtracting the total 12 week score from the respective trial participant's baseline score. Analysis of covariance will be used (Vickers and Altman 2001), group and ADT-status will be set as factors, the response will be change in FACT-P and covariates are age and baseline score. The results will be presented as least squares means (LSMEANS) differences between the two groups with 95 % confidence intervals and p-values.

Secondary outcomes including safety outcomes Changes from baseline to 6 month for LBM, BMC, BMD, and total body fat mass will be analysed in the same manner as the primary outcome.

QoL, Functional Well-Being and Physical Activity (based on MET values derived from the IPAQ questionnaire) measured at baseline, 12 weeks and 6 months will be analysed using a mixed model for repeated measurements. Changes from baseline to 12 weeks or 6 months will be treated as the response, the model will include fixed effects of factors: group, ADT, sampling time and their interactions, and the analysis will be adjusted for age and baseline value. The correlation between measurements on the same patient will be modeled using a random effect of patient.

Safety outcomes will be listed for each group and the number of fractures and falls that resulted in seeking medical assessment will be compared across groups using Fisher's exact test.

Subgroup analyses are planned to be reported for the patients treated with androgen deprivation therapy therefore results will be given both for the overall treatment effect and for subgroup obtained by stratifying level of according to androgen deprivation therapy. To verify the credibility of our subgroup analyses, we apply the criteria proposed by Sun and colleagues (Sun et al. 2012), i.e. the subgroup variable is a baseline characteristic, is a stratification factor, is specified a priori and includes only a small number of analyses.

Outline of figures and tables The first figure in the main publication will be a CONSORT flow diagram. The second figure will illustrate changes in the primary and secondary outcomes, except safety outcomes, at 12 weeks and 6 months, according to treatment group.

A third figure will display mean curves for the primary outcome for patients in different groups according to pattern of missing data. In particular, mean curves will be shown separately for completers and patients with missing data at one or more assessment times. The figure will be used to guide the type of sensitivity analyses performed to adjust results for a potentially deviating pattern for patients with incomplete observations.

Tables will be in following order; first a table delineating trial subjects characteristics, secondly a table showing changes in primary and secondary outcomes both at 12 weeks and 6 months. Thirdly safety outcomes will presented according to group and type.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with prostate cancer
* Age ≥18 years
* Able to read and understand questionnaires in Danish
* Signed informed consent

Exclusion Criteria:

* <6 weeks after prostatectomy
* Football training disencouraged by primary physician
* Osteoporosis (T-score < -2,5) assessed by Dual Energy X-Ray Absorptiometry at baseline

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Mean change in quality of life from baseline to week 12 | 12 weeks
  Assessed with Functional Assessment of Cancer Therapy - Prostate Questionaire

SECONDARY OUTCOMES:
Mean change in quality of life from baseline to month 6 | 6 months
  Assessed with Functional Assessment of Cancer Therapy - Prostate Questionaire
Whole-body bone mineral content percent change from baseline to month 6 | 6 months
  Assessed by dual energy x-ray absorptiometry.
Whole-body bone mineral density percent change from baseline to month 6 | 6 months
  Assessed by dual energy x-ray absorptiometry.
Whole-body lean body mass mean change from baseline to month 6 | 6 months
  Assessed by dual energy x-ray absorptiometry.
Whole-body fat mass mean change from baseline to month 6 | 6 months
  Assessed by dual energy x-ray absorptiometry.
Self-reported physical activity from baseline to week 12 and month 6 | 12 weeks and 6 months
  Assessed by the International Physical Activity Questionnaire
Self-reported functional well-being from baseline to week 12 and month 6 | 12 weeks and 6 months
  Assessed with Functional Assessment of Cancer Therapy - Prostate Questionaire, subscale functional well-being
Lumbar spine bone mineral density percent change from baseline to month 6 | 6 months
  Assessed by dual energy x-ray absorptiometry.
Femoral neck bone mineral density percent change from baseline to month 6 | 6 months
  Assessed by dual energy x-ray absorptiometry.
Total hip bone mineral density percent change from baseline to month 6 | 6 months
  Assessed by dual energy x-ray absorptiometry.
Number of participants with any fracture from baseline to month 6 | 6 months
  Any fracture includes fractures at any site excluding skull, facial, mandible, metacarpals, finger phalanges, and toe phalanges
Number of participants with falls that resulted in seeking medical assessment from baseline to month 6 | 6 months
  Any falls for which participants report to obtain medical treatment

OTHER OUTCOMES:
EQ-5D-5L for use in health economics analysis | 12 weeks and 6 months
Medical outcomes study 12-item short-form health survey(SF-12), version 2 for use in health economics analysis | 12 weeks and 6 months
Dyadic adjustment | 12 weeks and 6 months
  The seven-item version of the dyadic adjustment scale (DAS)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Midtgaard, Dr, Study Director — Rigshospitalet, Denmark; Eik D Bjerre, Msc., Principal Investigator — Rigshospitalet, Denmark
Locations (4):
- Denmark (4):
  - Aarhus University Hospital, Aarhus, Aarhus N
  - Rigshospitalet, Copenhagen, København N
  - Odense Universitets Hospital, Odense, Odense C
  - Sydvestjysk Sygehus, Esbjerg, Esbjerg

REFERENCES:
- [Background] Bjerre E, Bruun DM, Tolver A, Brasso K, Krustrup P, Johansen C, Christensen R, Rorth M, Midtgaard J. Effectiveness of community-based football compared to usual care in men with prostate cancer: Protocol for a randomised, controlled, parallel group, multicenter superiority trial (The FC Prostate Community Trial). BMC Cancer. 2016 Oct 3;16(1):767. doi: 10.1186/s12885-016-2805-0. PMID 27716218
- [Derived] Midtgaard J, Tjornhoj-Thomsen T, Rorth M, Kronborg M, Bjerre ED, Oliffe JL. Female partner experiences of prostate cancer patients' engagement with a community-based football intervention: a qualitative study. BMC Public Health. 2021 Jul 15;21(1):1398. doi: 10.1186/s12889-021-11448-7. PMID 34266389
- [Derived] Bjerre ED, Weller S, Poulsen MH, Madsen SS, Bjerre RD, Ostergren PB, Borre M, Brasso K, Midtgaard J. Safety and Effects of Football in Skeletal Metastatic Prostate Cancer: a Subgroup Analysis of the FC Prostate Community Randomised Controlled Trial. Sports Med Open. 2021 Apr 20;7(1):27. doi: 10.1186/s40798-021-00318-6. PMID 33877496
- [Derived] Bjerre ED, Petersen TH, Jorgensen AB, Johansen C, Krustrup P, Langdahl B, Poulsen MH, Madsen SS, Ostergren PB, Borre M, Rorth M, Brasso K, Midtgaard J. Community-based football in men with prostate cancer: 1-year follow-up on a pragmatic, multicentre randomised controlled trial. PLoS Med. 2019 Oct 1;16(10):e1002936. doi: 10.1371/journal.pmed.1002936. eCollection 2019 Oct. PMID 31574097
- [Derived] Bjerre ED, Brasso K, Jorgensen AB, Petersen TH, Eriksen AR, Tolver A, Christensen JF, Poulsen MH, Madsen SS, Ostergren PB, Borre M, Krustrup P, Johansen C, Rorth M, Midtgaard J. Football Compared with Usual Care in Men with Prostate Cancer (FC Prostate Community Trial): A Pragmatic Multicentre Randomized Controlled Trial. Sports Med. 2019 Jan;49(1):145-158. doi: 10.1007/s40279-018-1031-0. PMID 30506427
- See also: Study homepage — http://www.fcprostata.dk